CLINICAL TRIAL: NCT06138353
Title: Shuxuening Injection for the Prevention of Cerebral Vasospasm in Patients With Aneurysmal Subarachnoid Hemorrhage -- A Randomized, Double-blind, Placebo-parallel Controlled Clinical Trial
Brief Title: Shuxuening Injection for the Prevention of CVS in Patients With aSAH(SXN-CVS)
Acronym: SXN-CVS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaolin Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Xiaolin Chen, MD, Deputy Chief of Neurosurgery, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HX-A-2023023
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: aneurysmal subarachnoid hemorrhage; cerebral vasopasm; delayed cerebral ischemia; surgical clipping; coiling
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — shuxuening

STUDY DESIGN:
Intervention Model Description: Shuxuening injection treatment : Shuxuening injection (specification: 10ml/branch, Lanzhi Group Wanrong Pharmaceutical Co., Ltd.), 20 ml (2 branches) + 5% dextrose injection 250 ml, intravenously, once a day, from the first day of postoperative aSAH, treatment for 1 course of treatment, a total of 10-14 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure blinding, personnel involved in randomisation coding or with potential access to the blind base, doctors or nurses administering the medication, should not be involved in activities such as selection of subjects, evaluation of efficacy, and assessment of safety, so as not to introduce bias.
  In addition, to ensure blinding, the packaging and batch numbers of the drugs in both groups will be identical, and the packaging batch numbers will be uniformly labelled. Each box will be labelled with a unique drug ID number. This number will be used to designate the treatment received by the patient, but will not indicate treatment assignment to the investigator or the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shuxuening injection treatment group (Experimental): Group1: Shuxuening injection treatment group (N1=25): Shuxuening injection (specification: 10ml/branch, Lanzhi Group Wanrong Pharmaceutical Co., Ltd.), 20 ml (2 branches) + 5% dextrose injection 250 ml, intravenously, once a day, from the first day of postoperative, treatment for 1 course of treatment, a total of 10-14 days.
  Interventions: Drug: Shuxuening injection or placebo
- Placebo control group (Placebo Comparator): Group2: Placebo control group (N2=25): Shuxuening injection simulant (0.9% sodium chloride injection, specification: 10 ml/cartridge, Kunming Yusi Pharmaceutical Co., Ltd.), 20 ml (2 cartridges) + 5% dextrose injection 250 ml, intravenously dripped once a day, from the first day of postoperative, treatment for 1 course of treatment, for a total of 10-14 days.
  Interventions: Drug: Shuxuening injection or placebo

INTERVENTIONS:
Drug: Shuxuening injection or placebo — Shuxuening injection treatment group : Shuxuening injection (specification: 10ml/branch, Lanzhi Group Wanrong Pharmaceutical Co., Ltd.), 20 ml (2 branches) + 5% dextrose injection 250 ml, intravenously, once a day, from the first day of postoperative, treatment for 1 course of treatment, a total of 10-14 days.

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a frequent worldwide cause for stroke with a mortality of around 30%. Worldwide, almost 500 000 patients have aneurysmal SAH annually.An incidence of 2-16 cases of spontaneous SAH per 100 000 person-years was reported in a recent meta-analysis .

Surgical treatment of aneurysms is essential in the acute phase of aSAH patients, either by surgical clipping or by endovascular embolization. Although there are many factors that influence the prognosis of patients with aSAH, cerebral vasospasm (CVS) and delayed cerebral ischemia (DCI) are the main factors contributing to the high mortality rate (30-40% within 30 days) and poor long-term functional prognosis of patients after aSAH. Cerebral vasospasm (CVS) is defined as focal or diffuse temporary narrowing of vessel diameter due to contraction of smooth muscle in the arterial wall, which can be detected by digital subtraction angiography (DSA), transcranial ultrasound Doppler (TCD), magnetic resonance (MR), and CT angiography (CTA) or visualised during intraoperative.The prevalence of CVS after aSAH is 67% , with symptomatic patients (symptomatic vasospasm) in 30-40% of them and leading to ischaemic events in 10-45% of patients. It usually begins 3-4 days after bleeding, peaks at 7-10 days and finally resolves at around 14-21 days.

There is no effective treatment to prevent cerebral vasospasm events.Shuxuening Injection is a sterilized aqueous solution made by extraction of Ginkgo biloba. The study aims to clarify the clinical study of the efficacy and safety of Shuxuening Injection (10ml/branch) for the prophylactic of cerebral vasospasm (CVS) after aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-parallel controlled clinical trial.

Patients were randomly divided into 2 groups according to 1:1. Group1: Shuxuening injection treatment group (N1=25): Shuxuening injection (specification: 10ml/branch, Lonch Group Wanrong Pharmaceutical Co., Ltd.), 20 ml (2 branches) + 5% dextrose injection 250 ml, intravenously, once a day, from the first day of postoperative, treatment for 1 course of treatment, a total of 10-14 days; Group2: Placebo control group (N2=25): Shuxuening injection simulant (0.9% sodium chloride injection, specification: 10ml/cartridge, Kunming Yusi Pharmaceutical Co., Ltd.), 20 ml (2 cartridges) + 5% dextrose injection 250 ml, intravenously once a day, from the first day of postoperative, treatment for 1 course of treatment, for a total of 10-14 days; both groups received the basal treatment.

Basic treatment included nimodipine (oral nimodipine, 60 mg, 4 hours/dose), oxygen inhalation,blood pressure and cardiac monitoring, fluid balance and blood glucose management, etc., in accordance with the "2023 American Heart Association/American Stroke Association (AHA/ASA) Guidelines for the Management of Patients with Aneurysmal Subarachnoid Haemorrhage". Patients will be classified according to the Hunt-Hess grade, with H-H I-II grade placed in the general ward and III-V grade placed in the intensive care unit(ICU).

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (> 18 years of age)
2. patients who were diagnosed with aneurysmal subarachnoid hemorrhage
3. the aneurysms were treated by microsurgery clipping or endovascular coiling
4. Time from onset to surgery is less than or equal to 72 hours;
5. no new hemorrhage or new infarction on first postoperative CT;
6. signed informed consent.

Exclusion Criteria:

1. mRS >1 before onset
2. history of microsurgery clipping or endovascular coiling
3. anemia (hemoglobin <10g/dL), thrombocytopenia (platelet count <100×10^9/L), or leukopenia (white blood cell count <3×10^9/L) at randomization
4. patients with chronic liver and kidney dysfunction (including those with alanine aminotransferase (ALT) and aliquot aminotransferase (AST) > 3 times the upper limit of normal, and those with blood creatinine (Scr) > 2 times the upper limit of normal)
5. patients suffering from cardiorespiratory insufficiency disease such as heart failure, severe heart disease, respiratory failure
6. allergy to Shuxuening Injection
7. those who have used Shuxuening Injection before enrolled
8. patients with end-stage disease, those with a life expectancy of less than 3 months
9. women who are prepare for pregnancy in 3 months, pregnant or breastfeeding
10. those who are participating or have participated in other clinical trials within the past 1 month
11. patients are unable to comply with this study due to mental illness, cognitive or emotional disorders, etc. or that the investigator think patients inappropriate for this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with cerebral vasospasm(CVS) | Cerebral vasospasm events within 14 days
  The prevalence of CVS after aSAH is 67% , with symptomatic patients (symptomatic vasospasm) in 30-40% of them and leading to ischemic events in 10-45% of patients. It usually begins 3-4 days after rupture bleeding, peaks at 7-10 days and finally resolves at around 14-21 days.

SECONDARY OUTCOMES:
Rate of Delayed Cerebral Ischemic(DCI) | Delayed cerebral ischemic events within 14 days
  Delayed cerebral ischemic events within 14 days

OTHER OUTCOMES:
modified Rankin scale(mRS) | modified Rankin scale(mRS) within 14 days and 90 days
  modified Rankin scale(mRS) ranged from a minimum of 0 to a maximum of 5, with higher scores representing a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
we do not share IPD.

REFERENCES:
- [Result] Dankbaar JW, de Rooij NK, Velthuis BK, Frijns CJ, Rinkel GJ, van der Schaaf IC. Diagnosing delayed cerebral ischemia with different CT modalities in patients with subarachnoid hemorrhage with clinical deterioration. Stroke. 2009 Nov;40(11):3493-8. doi: 10.1161/STROKEAHA.109.559013. Epub 2009 Sep 17. PMID 19762703
- [Result] Macdonald RL, Schweizer TA. Spontaneous subarachnoid haemorrhage. Lancet. 2017 Feb 11;389(10069):655-666. doi: 10.1016/S0140-6736(16)30668-7. Epub 2016 Sep 13. PMID 27637674
- [Result] Westermaier T, Jauss A, Eriskat J, Kunze E, Roosen K. Acute vasoconstriction: decrease and recovery of cerebral blood flow after various intensities of experimental subarachnoid hemorrhage in rats. J Neurosurg. 2009 May;110(5):996-1002. doi: 10.3171/2008.8.JNS08591. PMID 19061352
- [Result] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Result] Geraghty JR, Testai FD. Delayed Cerebral Ischemia after Subarachnoid Hemorrhage: Beyond Vasospasm and Towards a Multifactorial Pathophysiology. Curr Atheroscler Rep. 2017 Oct 23;19(12):50. doi: 10.1007/s11883-017-0690-x. PMID 29063300
- [Result] Macdonald RL. Delayed neurological deterioration after subarachnoid haemorrhage. Nat Rev Neurol. 2014 Jan;10(1):44-58. doi: 10.1038/nrneurol.2013.246. Epub 2013 Dec 10. PMID 24323051
- [Result] Mahadevan S, Park Y. Multifaceted therapeutic benefits of Ginkgo biloba L.: chemistry, efficacy, safety, and uses. J Food Sci. 2008 Jan;73(1):R14-9. doi: 10.1111/j.1750-3841.2007.00597.x. PMID 18211362
- [Result] Calapai G, Crupi A, Firenzuoli F, Marciano MC, Squadrito F, Inferrera G, Parisi A, Rizzo A, Crisafulli C, Fiore A, Caputi AP. Neuroprotective effects of Ginkgo biloba extract in brain ischemia are mediated by inhibition of nitric oxide synthesis. Life Sci. 2000 Oct 20;67(22):2673-83. doi: 10.1016/s0024-3205(00)00858-4. PMID 11105983
- [Result] Tulsulkar J, Shah ZA. Ginkgo biloba prevents transient global ischemia-induced delayed hippocampal neuronal death through antioxidant and anti-inflammatory mechanism. Neurochem Int. 2013 Jan;62(2):189-97. doi: 10.1016/j.neuint.2012.11.017. Epub 2012 Dec 7. PMID 23228346